CLINICAL TRIAL: NCT01709201
Title: Reducing Problematic Substance Use in Youth With Chronic Medical Conditions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not receive funding and was administratively withdrawn.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sharon Levy, Assistant Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FP01009751
Record Dates: First submitted 2012-10-15; First posted 2012-10-18 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Alcohol Abuse; Drug Abuse
Keywords: Alcohol abuse; Drug abuse; Diabetes Mellitus; Persistent Asthma; Juvenile Arthritis; Ulcerative Colitis
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Diabetes Mellitus; Arthritis, Juvenile; Colitis, Ulcerative | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (No Intervention): Those in the Treatment as Usual group will not receive the brief intervention for substance use but will receive a brief health education brochure.
- Brief Intervention (Experimental): Those in the Brief Intervention group will receive a brief motivational intervention aimed at encouraging the participant to decrease their substance use.
  Interventions: Behavioral: Brief Intervention

INTERVENTIONS:
Behavioral: Brief Intervention — Those in the intervention arm will undergo a 10-minute discussion with a trained interventionist aimed at encouraging decreased substance use.
  Arms: Brief Intervention

SUMMARY:
The investigators goal is to pilot a substance use-related brief intervention (BI) for youth with chronic medical conditions, obtaining preliminary evidence of feasibility, acceptability and impacts of the approach for reducing substance use among this group.

ELIGIBILITY:
Inclusion Criteria:

* 14-18 years old
* Currently being treated for diabetes, rheumatologic disorders, asthma, or ulcerative colitis (UC) at Boston Children's Hospital with a duration of chronic illness of at least one year
* Previous participation in the screening validation study
* Evidence of problems related to substance use

Exclusion Criteria:

* Medically or emotionally unstable or otherwise unable to provide assent/consent
* Unable to speak/read English
* Unable to use a computer keyboard and/or complete an interviewer-assisted questionnaire

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Percent days abstinent | 30 days post baseline
  We will compare the percent days abstinent from substances between the Treatment as Usual and Intervention groups 30 days post baseline

SECONDARY OUTCOMES:
Medical complications | 30 days post baseline
  We will evaluate the incidents of disease complications between the Treatment as Usual and Intervention groups 30 days post baseline

OTHER OUTCOMES:
Percent Days Abstinent 90 days post baseline | 90 days post baseline
  We will compare the percent days abstinent from substances between the Treatment as Usual and Intervention groups 90 days post baseline
Medical complications 90 days post baseline | 90 days post baseline
  We will evaluate the incidents of disease complications between the Treatment as Usual and Intervention groups 30 days post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Levy, MD, MPH, Principal Investigator — Boston Children's Hospital; Elissa Weitzman, ScD, MSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States